CLINICAL TRIAL: NCT00019071
Title: A PHASE I STUDY OF 2-CHLORODEOXYADENOSINE AND RADIATION FOR THE TREATMENT OF HIGH GRADE GLIOMA (CDX)
Brief Title: Chemotherapy Followed by Radiation Therapy in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064153; NCI-95-C-0092A; NCI-95-C-0092; NCT00001433 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2004-04-05 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2002-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Drug Therapy; Cladribine; Radiotherapy

INTERVENTIONS:
Drug: chemotherapy
Drug: cladribine
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of cladribine followed by radiation therapy in treating patients who have malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of cladribine in combination with radiotherapy in patients with high grade glioma. II. Assess this regimen in terms of toxicity and survival in these patients. III. Assess the acute neurotoxicity of continuous infusion cladribine in these patients. IV. Assess this regimen in terms of response, local control, and time to progression in these patients. V. Define a dose level of cladribine associated with potentiation of acute and/or delayed radiation toxicity (radiosensitizing dose level).

OUTLINE: This is a dose escalation study of cladribine. Patients receive cladribine by continuous IV infusion 5 days a week for 4 weeks and undergo radiotherapy twice a day, beginning 3 hours after initiation of cladribine, 5 days a week for 4.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of cladribine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed at 1 month, then every 3 months thereafter for survival.

PROJECTED ACCRUAL: A total of 12-42 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven high-grade glioma confined to 1 or both hemispheres of the brain and including: Grade III astrocytoma (anaplastic astrocytoma) Grade IV astrocytoma (glioblastoma multiforme) ineligible for NCI-95-C-0069 protocol Histologic confirmation of high-grade astrocytoma by NIH neuropathology division required (including mandatory review of slides from biopsy or resection) No evidence of metastatic or leptomeningeal spread

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 60-100% ECOG 0-2 Life expectancy: Greater than 6 months Hematopoietic: WBC at least 3,500/mm3 Absolute granulocyte count at least 900/mm3 Absolute leukocyte count at least 900/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Liver function tests no greater than 2.5 times upper limit of normal Renal: Creatinine clearance at least 95 mL/min Creatinine no greater than 1.3 mg/dL Other: No history of psychiatric disease that would prevent compliance No other malignancy within the past 5 years except: Basal cell carcinoma of the skin Carcinoma in situ of the cervix Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No systemic chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior cranial radiotherapy Surgery: No more than 3 months since surgery (biopsy; subtotal or near-total resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-03

CONTACTS AND LOCATIONS:
Overall Officials: C. Norman Coleman, MD, Study Chair — NCI - Radiation Oncology Branch; ROB
Locations (1):
- Radiation Oncology Branch, Bethesda, Maryland, United States